CLINICAL TRIAL: NCT01234441
Title: Intradialytic Protein Supplementation & Exercise Training in Dialysis Patients.
Brief Title: Intra Hemodialytic Oral Protein and Exercise (IHOPE)
Acronym: IHOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kenneth Wilund, Prinicipal Responsiple Investigator, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01DK084016-01 (NIH)
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Proteins; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Sham Comparator): This group of patients will receive a non-nutritive beverage, and no exercise.
  Interventions: Dietary Supplement: Control
- Protein (Active Comparator): This group of patients will ingest 30 grams of a liquid whey protein supplement during the first hour of their dialysis session
  Interventions: Dietary Supplement: Protein
- Protein + Exercise (Active Comparator): This group will ingest 30 grams of a liquid whey protein supplement as well as exercise for 30-45 minutes during their dialysis treatment
  Interventions: Behavioral: Protein + Exercise

INTERVENTIONS:
Dietary Supplement: Control — A placebo non-nutritive beverage will be administered before dialysis sessions 3 times per week.
  Arms: Control
Dietary Supplement: Protein — A whey protein beverage will be administered before dialysis sessions 3 times per week.
  Arms: Protein
Behavioral: Protein + Exercise — A whey protein beverage will be administered before dialysis sessions 3 times per week. Patients will also exercise by stationary bicycle during dialysis sessions 3 times per week.
  Arms: Protein + Exercise

SUMMARY:
Chronic kidney disease (CKD) patients receiving hemodialysis treatment (CKD stage 5) suffer from a variety of co-morbid diseases, many of which may be mechanistically linked. Protein malnutrition, muscle catabolism and wasting are especially common, and these lead to reduced muscle strength, declines in physical function, and low levels of physical activity. Physical inactivity exacerbates these functional declines, and also promotes cardiovascular disease (CVD) and bone disorders. This cycle of disease and disability greatly reduces quality of life (QOL) and increases mortality rates in dialysis patients.

Many factors contribute to the development of these co-morbidities. Chronic inflammation is believed to be a cause and a consequence of the protein malnutrition, CVD and bone disorders in dialysis patients. In addition, abnormalities in mineral metabolism resulting from the deficit in kidney function promote the loss of mineral from bone and the deposition of mineral in the vasculature, a process termed vascular calcification (VC). VC is associated with a variety of CVD-related disorders, including arterial stiffness, increases in arterial wall intima-media thickness (IMT), left ventricular hypertrophy (LVH), and declines in cardiac function. As a result of these abnormalities, cardiovascular events are 10 to 30 times greater in dialysis patients than in age- and sex-matched subjects in the general population.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) patients receiving hemodialysis treatment (CKD stage 5) suffer from a variety of co-morbid diseases, many of which may be mechanistically linked. Protein malnutrition, muscle catabolism and wasting are especially common, and these lead to reduced muscle strength, declines in physical function, and low levels of physical activity. Physical inactivity exacerbates these functional declines, and also promotes cardiovascular disease (CVD) and bone disorders. This cycle of disease and disability greatly reduces quality of life (QOL) and increases mortality rates in dialysis patients.

Many factors contribute to the development of these co-morbidities. Chronic inflammation is believed to be a cause and a consequence of the protein malnutrition, CVD and bone disorders in dialysis patients. In addition, abnormalities in mineral metabolism resulting from the deficit in kidney function promote the loss of mineral from bone and the deposition of mineral in the vasculature, a process termed vascular calcification (VC). VC is associated with a variety of CVD-related disorders, including arterial stiffness, increases in arterial wall intima-media thickness (IMT), left ventricular hypertrophy (LVH), and declines in cardiac function. As a result of these abnormalities, cardiovascular events are 10 to 30 times greater in dialysis patients than in age- and sex-matched subjects in the general population.

A variety of pharmacological therapies are commonly used to help prevent or attenuate the progression of CKD co-morbidities; however, morbidity and mortality in this population remain extremely high, indicating that additional therapeutic strategies that may improve the health and QOL in this population are needed. Recently, the National Kidney Foundation recommended that dialysis patients increase their protein intake to 1.2 g/kg/day to help prevent protein malnutrition; however, little is known about the efficacy of this recommendation. Intradialytic (during dialysis) protein supplementation has been shown to increase serum albumin levels11, and also increases amino acid uptake into skeletal muscle, an effect that is potentiated by both resistance and endurance exercise. However, the individual and combined effects of intradialytic protein supplementation and exercise training on lean mass, muscle strength, and physical function is unknown. Furthermore, intradialytic protein supplementation and exercise training improve many risk factors associated with CVD and renal bone disease (e.g., plasma lipids, inflammatory variables), but their effect on functional CVD outcomes (e.g., arterial stiffness, VC, IMT, LVH, myocardial performance) and bone health in dialysis patients is unknown.

The primary objective of the proposed research is to evaluate the efficacy of intradialytic oral protein supplementation, with and without concomitant intradialytic endurance exercise training (cycling), on physical function, CVD risk, and bone health. We will also examine potential mechanisms for these effects, and determine if improvements in these factors lead to improvements in QOL. Hemodialysis patients will be randomized to the following groups for 12 months: 1) usual care/control (CON); 2) intradialytic protein supplementation (PRO); or 3) intradialytic protein supplementation + exercise training (PRO+EX).

Primary Aim #1: Examine the effects of intradialytic oral protein supplementation and exercise training on physical function.

Hypothesis #1: Physical function, as assessed by a shuttle walk test, will improve in PRO+EX and PRO, compared to CON, and the magnitude of improvements will be greatest in PRO+EX. In secondary analyses, we also will examine the effects of our interventions on other variables related to physical function, including lean body mass, muscle strength, and activities of daily living (ADL) assessments.

Primary Aim #2: Examine the effects of intradialytic oral protein supplementation and exercise training on CVD risk.

Hypothesis #2: CVD risk, as assessed by carotid artery stiffness, will improve in PRO+EX and PRO, compared to CON, and the magnitude of improvements will be greatest in PRO+EX. In secondary analyses, we also will examine the effects of our interventions on other factors related to CVD risk, including carotid IMT, myocardial performance, LVH, aortic calcification, and epicardial fat levels.

Primary Aim #3: Examine the effects of intradialytic oral protein supplementation and exercise training on bone health as determined by bone mineral density (BMD).

Hypothesis #3: BMD will be reduced significantly more in CON than in PRO+EX or PRO. We anticipate that BMD will remain stable in PRO+EX or PRO. Because the exercise is not bone loading (i.e., invoking ground or joint reaction forces), we do not expect additive effects of PRO+EX on BMD.

ELIGIBILITY:
Inclusion Criteria:

* Must receive hemodialysis treatment at least 3 days per week.
* Must be ≥ 30 years of age.
* Must be willing to be randomized to the control or intervention groups.
* Must be physically able to exercise (e.g., no orthopedic problems that would preclude them from cycling during dialysis).
* Must receive medical clearance from their primary care physician to participate.
* Must be on phosphate binders to control calcium levels.

Exclusion Criteria:

* Persistent hemoglobin levels < 10g/dl.
* Weight greater than 300 pounds.
* Currently receiving any form of intradialytic protein supplementation (oral, enteral, or parenteral) or participating in any form of intradialytic exercise training.
* Chronic obstructive pulmonary disease (COPD) and decompensated chronic heart failure (CHF).
* On dialysis treatment for < 3 months (or enrollment may be postponed).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Examine the effects of intradialytic oral protein supplementation and exercise training on physical function. | 12 months
  Physical function, as assessed by a shuttle walk test, will improve in PRO+EX and PRO, compared to CON, and the magnitude of improvements will be greatest in PRO+EX. In secondary analyses, we also will examine the effects of our interventions on other variables related to physical function, including lean body mass, muscle strength, and activities of daily living (ADL) assessments.

SECONDARY OUTCOMES:
Examine the effects of intradialytic oral protein supplementation and exercise training on CVD risk. | 12 months
  CVD risk, as assessed by carotid artery stiffness, will improve in PRO+EX and PRO, compared to CON, and the magnitude of improvements will be greatest in PRO+EX. In secondary analyses, we also will examine the effects of our interventions on other factors related to CVD risk, including carotid IMT, myocardial performance, LVH, aortic calcification, and epicardial fat levels.
Examine the effects of intradialytic oral protein supplementation and exercise training on bone health as determined by bone mineral density (BMD). | 12 months
  BMD will be reduced significantly more in CON than in PRO+EX or PRO. We anticipate that BMD will remain stable in PRO+EX or PRO. Because the exercise is not bone loading (i.e., invoking ground or joint reaction forces), we do not expect additive effects of PRO+EX on BMD.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Wilund, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Illinois at Urbana-Champaign, Urbana, Illinois

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133